CLINICAL TRIAL: NCT05701592
Title: Assessment of Outcomes of Double-bundle Posterior Cruciate Ligament Reconstruction (DB-PCLR)
Status: Recruiting | Type: Observational
Sponsor: Konrad Malinowski MD (Other)
Responsible Party: Sponsor-Investigator, Konrad Malinowski MD, Konrad Malinowski MD, Director of Artromedical Konrad Malinowski Clinic and Principal Investigator, Artromedical Konrad Malinowski Clinic
Organization: Artromedical Konrad Malinowski Clinic (Other)
Other Study IDs: 2-pro-ar-2023
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Posterior Cruciate Ligament Tear

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PCL tear treated with DB-PCLR: Patients with PCL tear treated with DB-PCLR
  Interventions: Procedure: DB-PCLR

INTERVENTIONS:
Procedure: DB-PCLR — DB-PCLR with reconstruction of both PCL bundles: anterolateral and posteromedial bundle will be performed.

SUMMARY:
Double-bundle Posterior Cruciate Ligament Reconstruction (DB-PCLR) is becoming increasingly used alternative to the single-bungle PCLR. While more technically challenging, it seems to better improve patients' outcomes. Therefore, outcomes of DB-PCLR will be assessed and reported.

ELIGIBILITY:
Inclusion Criteria:

* PCL tear with III grade sympomatic posterior instability confirmed clinically and radiologically
* full knee range of motion

Exclusion Criteria:

* active knee inflammation
* non-adherence to the study protocol
* fixed posterior drawer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after PCL tear with knee instability undergoing DB-PCLR
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee posterior translatory stability - posterior sag test | At the 12 month of the follow-up.
  Posterior sag test will be performed and outcome will be presented as present/ absent
Knee posterior translatory stability - posterior drawer test | At the 12 month of the follow-up.
  Posterior drawer test aided with Rollimeter will be performed and outcomes will be presented in milimeters
Knee posterior translatory stability - posterior Lachman test | At the 12 month of the follow-up.
  Posterior Lachman test aided with Rollimeter will be performed and outcomes will be presented in milimeters
Knee posterior translatory stability - stress X-ray | At the 12 month of the follow-up.
  Stress X-ray assessing posterior translatory stability of the knee will be performed and outcomes will be presented in milimeters
Knee internal rotation stability | At the 12 month of the follow-up.
  Maximal knee internal rotation angle will be assessed with different angles of knee flexion and measured by the means of goniometer and outcomes will be presented in degrees
Knee posterior translatory stability - posterior sag test | At the 24 month of the follow-up.
  Posterior sag test will be performed and outcome will be presented as present/ absent
Knee posterior translatory stability - posterior drawer test | At the 24 month of the follow-up.
  Posterior drawer test aided with Rollimeter will be performed and outcomes will be presented in milimeters
Knee posterior translatory stability - posterior Lachman test | At the 24 month of the follow-up.
  Posterior Lachman test aided with Rollimeter will be performed and outcomes will be presented in milimeters
Knee posterior translatory stability - stress X-ray | At the 24 month of the follow-up.
  Stress X-ray assessing posterior translatory stability of the knee will be performed and outcomes will be presented in milimeters
Knee internal rotation stability | At the 24 month of the follow-up.
  Maximal knee internal rotation angle will be assessed with different angles of knee flexion and measured by the means of goniometer and outcomes will be presented in degrees

SECONDARY OUTCOMES:
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 12 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 24 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score (KOOS) | At the 12 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score (KOOS) | At the 24 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
Retear rate | At the 12 month of the follow-up.
  Rate of patients with retear of the reconstructed ligament
Retear rate | At the 24 month of the follow-up.
  Rate of patients with retear of the reconstructed ligament
ROM | At the 12 month of the follow-up.
  Knee range of motion assessed by the means of goniometer.
ROM | At the 24 month of the follow-up.
  Knee range of motion assessed by the means of goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Konrad Malinowski, MD PhD, Principal Investigator — Artromedical Orthopaedic Clinic, Bełchatów, Poland
Locations (1):
- Artromedical Orthopaedic Clinic, Bełchatów, Łódź Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chahla J, Moatshe G, Cinque ME, Dornan GJ, Mitchell JJ, Ridley TJ, LaPrade RF. Single-Bundle and Double-Bundle Posterior Cruciate Ligament Reconstructions: A Systematic Review and Meta-analysis of 441 Patients at a Minimum 2 Years' Follow-up. Arthroscopy. 2017 Nov;33(11):2066-2080. doi: 10.1016/j.arthro.2017.06.049. Epub 2017 Aug 31. PMID 28866340
- [Background] Knapik DM, Gopinatth V, Jackson GR, Chahla J, Smith MV, Matava MJ, Brophy RH. Global variation in isolated posterior cruciate ligament reconstruction. J Exp Orthop. 2022 Oct 9;9(1):104. doi: 10.1186/s40634-022-00541-4. PMID 36209443
- [Background] LaPrade RF, Cinque ME, Dornan GJ, DePhillipo NN, Geeslin AG, Moatshe G, Chahla J. Double-Bundle Posterior Cruciate Ligament Reconstruction in 100 Patients at a Mean 3 Years' Follow-up: Outcomes Were Comparable to Anterior Cruciate Ligament Reconstructions. Am J Sports Med. 2018 Jul;46(8):1809-1818. doi: 10.1177/0363546517750855. PMID 29953296
- [Background] Bernhardson AS, DePhillipo NN, Aman ZS, Kennedy MI, Dornan GJ, LaPrade RF. Decreased Posterior Tibial Slope Does Not Affect Postoperative Posterior Knee Laxity After Double-Bundle Posterior Cruciate Ligament Reconstruction. Am J Sports Med. 2019 Feb;47(2):318-323. doi: 10.1177/0363546518819786. Epub 2019 Jan 18. PMID 30657698